CLINICAL TRIAL: NCT04300673
Title: Radio Guided Lymph Node Dissection in Oligometastatic Prostate Cancer Patients
Acronym: DETECT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-5805; 2019-003284-21 (EudraCT Number)
Record Dates: First submitted 2020-02-17; First posted 2020-03-09 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer; Lymph Node Metastases
Keywords: pelvic lymph node dissection (PLND); PSMA I&T; radio guided surgery (RGS)
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — PITX2 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Intervention: radio guided surgery
  Interventions: Procedure: Radio guided surgery (RGS) using Indium-labelled PSMA

INTERVENTIONS:
Procedure: Radio guided surgery (RGS) using Indium-labelled PSMA — Approximately 24hours prior to surgery (PLND) patients receive a radiolabelled PSMA-tracer. During surgery, urologists will use a gamma-probe to detect PSMA-postitive tumour depostitions in pelvic lymph nodes.

SUMMARY:
The study is a prospective, single arm phase I/II study. The primary aim of this study is to evaluate the feasibility of 111In-PSMA I&T radio guided surgery in patients diagnosed with prostate cancer who are highly suspected of having one or more pelvic lymph node metastases based on pre-operative imaging.

Patients with prostate cancer who have a high risk of lymph node metastases based on PSMA PET/CT and scheduled for robot-assisted PLND (with or without prostatectomy) will be recruited. Eligible patients will receive an additional ferumoxtran-10 enhanced MRI to complement pre-operative imaging. Twenty-four hours before surgery, patients will receive the radiolabelled PSMA tracer. Pelvic Lymph node dissections are carried out according to standard of care procedures. During surgery, the surgeon will be provided with a gamma-probe to detect PSMA expressing lymph nodes in vivo. Dissected samples will be systematically assessed on tracer accumulation using the gamma-probe ex vivo. After surgery, the samples will be scanned in the small animal SPECT/CT and 7T-MRI. After scanning, samples will be presented to pathologists for pathological analysis according to standard of care including staining for PSMA expression. At 3 months after surgery, patients will undergo a PSMA-PET/CT. Up until one year after surgery patients will be followed according to standard of care-guidelines by 3-monthly serum-PSA measurements.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer of the prostate, based on prostate biopsy-core analysis.
* At least one 18F/68Ga-PSMA-PET/CT suspected positive metastasis in lymph nodes, located in the pelvic region.
* Patient is scheduled and fit for robot assisted surgery (PLND or radical prostatectomy +PLND).
* Patient is suitable for PLND (and radical prostatectomy) conform institutional guidelines and is not yet treated pre-operatively .
* Age≥50 years.
* Ability to give voluntary written informed consent to participate in this study.

Exclusion Criteria:

* No detectable lesion on the 18F/68Ga-PSMA-PET/CT with an uptake level above liver uptake level (reference).
* Patients who are not scheduled for robot-assisted PLND.
* Prior pelvic surgery(1)
* Unequivocal evidence of metastases outside the pelvic region.
* Presence of any medical condition that in the opinion of the investigator/treating physician will affect patients' clinical status by participating in this trial.
* Prior prostate cancer treatment(2).
* Contraindication for MRI-scanning, i.e. claustrophobia, intracranial metal clips, metallic bodies in the eye, implanted electric and electronic devices not eligible for MRI (pacemakers, insulin pumps, cochlear implants, neurostimulators).
* Inability to lie still for at least 60 minutes or comply with imaging.
* Contraindication for iron infusion or hypersensitivity/allergy to the active substance or any of the excipients.
* The patient is already enrolled in one or more concurrent studies, which could confound the results of this study, according to the investigators.

  1. Pelvic surgery is defined as "any surgery associated with pelvic lymphadenopathy'.
  2. Prior prostate cancer treatment is defined as prostate and/or pelvic radiotherapy, hormonal treatments such as androgen deprivation therapy, prostate brachytherapy, prostate cryotherapy, high intensity focused ultrasound (HIFU) and/or prostate electroporation.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study concerns prostate cancer patients.
Enrollment: 20 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of 111In-PSMA-I&T radio guided surgery | 1 year
  The primary aim of this study is to evaluate the feasibility of 111In-PSMA-I&T radio guided surgery in patients diagnosed with prostate cancer who are highly suspected of having one or more pelvic lymph node metastasis/metastases based on pre-operative imaging. Feasibility will be defined as the ability to intra-operatively detect the lymph nodes (using a gamma probe) which were pre-operatively identified on PSMA-PET/CT

SECONDARY OUTCOMES:
The accuracy of 111In-PSMA-I&T radio guided surgery | 1 year
  Accuracy will be expressed as sensitivity and specificity percentage. Test results of gamma probe (positive or negative) will be compared with histopathology (gold standard) (positive or negative: i.e. containing PSMA-expressing prostate cancer cells).
The safety of 111In-PSMA-I&T | 1 year
  Safety will be assesed by the number of participants with treatment related adverse events as assessed by CTCAE v4.0. For this outcome measure extra bloodsampling is included in the study protocol.
Dosimetry of 111In-PSMA-I&T | 1 year
  Blood-clearance ratios will be determined based on radiation dosimetry as assessed by bloodsampling at set time points after injection.
Correlation between tracer accumulation and lymph node size, PSMA-staining and SUV on PSMA-PET/CT | 1 year
Correlation between post-operative nano-MRI and SPECT | 1 year
Correlation between pre-operative imaging and postoperative imaging | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Sedelaar, MD, PhD, Principal Investigator — Radboudumc Nijmegen
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Canisius Wilhelimina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schilham MGM, Somford DM, Kusters-Vandevelde HVN, Hermsen R, van Basten JPA, Hoekstra RJ, Scheenen TWJ, Gotthardt M, Sedelaar JPM, Rijpkema M. Prostate-Specific Membrane Antigen-Targeted Radioguided Pelvic Lymph Node Dissection in Newly Diagnosed Prostate Cancer Patients with a Suspicion of Locoregional Lymph Node Metastases: The DETECT Trial. J Nucl Med. 2024 Mar 1;65(3):423-429. doi: 10.2967/jnumed.123.266495. PMID 38176721